CLINICAL TRIAL: NCT00346437
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Ad5FGF-4 in Patients With Stable Angina
Brief Title: Efficacy and Safety of Intracoronary Ad5FGF-4 in Patients With Stable Angina (AGENT-3)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cardium Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 304386
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2008-11

CONDITIONS: Angina Pectoris
Keywords: angina; FGF-4; angiogenesis; adenovector; growth factor; myocardial ischemia; revascularization
MeSH Terms: conditions — Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Ad5FGF-4
  Interventions: Genetic: Ad5FGF-4 vs. Placebo
- 2 (Experimental): Ad5FGF-4
  Interventions: Genetic: Ad5FGF-4 vs. Placebo
- 3 (Placebo Comparator): Placebo
  Interventions: Genetic: Ad5FGF-4 vs. Placebo

INTERVENTIONS:
Genetic: Ad5FGF-4 vs. Placebo — Intracoronary infusion

SUMMARY:
The purpose of this study is to determine whether a single intracoronary infusion of Ad5FGF-4 is effective in improving exercise capacity measured by exercise treadmill testing, angina functional class, patient symptoms, quality of life, and cardiovascular outcomes. Two doses will be studied, 2.87 x 10(8) and 2.87 x 10(9) viral particles, to evaluate the dose-response of Ad5FGF-4. Short-term and long-term safety of Ad5FGF-4 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-75 years, male or female, with coronary artery disease
* Patients over 50 years of age agree to undergo sigmoidoscopy, unless they have undergone such an exam or colonoscopy within the preceding 36 months with negative findings
* CCS angina Class 2 to 4
* Stable angina for =>4 weeks despite antianginal drug treatment, and who are able to exercise for at least 3 minutes but no more than 10 minutes on the first qualifying baseline ETT and no more than 12 minutes on the last qualifying baseline ETT using the modified Balke exercise protocol
* LVEF =>30% by echocardiography, LV angiogram, or a MUGA scan undertaken within the preceding 12 months
* Classic angina or angina equivalent associated with =>1mm ST segment depression (horizontal or down sloping) at least in the first qualifying ETT. The variability in exercise duration (time to grade 3/4 angina or angina equivalent) does not vary by > 20% in 2 consecutive tests
* Single, double, or triple vessel coronary artery disease. Patients with 3 vessel disease should have at least 1 proximal major vessel or graft with <70% stenosis
* Patients who do not require immediate PTCA or CABG surgery
* Provided written informed consent

Exclusion Criteria:

* Unstable angina
* CCS Class 1 angina
* Patients in whom ECG evidence of exercise induced myocardial ischemia is difficult to detect
* Intercurrent illness which may interfere with the ability to perform the ETT
* Untreated life-threatening ventricular arrhythmias
* Left main coronary artery stenosis =>70%, unless bypassed with a patent graft
* Coronary artery bypass surgery within the past 6 months, unless those grafts are closed
* In situ arterial CABG other than the RIMA or LIMA, unless it is 100% occluded
* Myocardial infarction within the last 8 weeks
* CHF (NYHA class IV) despite treatment
* Angioplasty within the previous 6 months
* Prior transmyocardial laser revascularization
* Enhanced external counterpulsation (EECP) within 12 weeks prior to study entry
* Coronary ostial stenosis that precludes adequate catheter engagement in any target vessel
* Coronary artery to venous communications which bypass the coronary capillary bed
* Heparin associated thrombocytopenia (HIT)
* Moderate to severe nonproliferative or proliferative retinopathy from any cause (ETDRS Score > 35), clinically significant macular edema, or previous panretinal photocoagulation therapy
* History of malignant neoplasms (except superficial basal cell skin carcinoma) within the past 10 years
* Malignant tumors or abnormal cancer screening tests suspicious for cancer, or patients in whom screening exams indicate possible occult malignancy, unless malignancy has been ruled out
* Family history of colon cancer in any first-degree relative, unless the patient has undergone a colonoscopy within the past 12 months with negative findings
* Elevated PSA level (unless prostate cancer has been excluded)
* HIV positive
* Hepatic disease or those who are positive for hepatitis B or C, or whose SGPT is > 2 times the upper limit of normal range, or whose serum bilirubin is > 2 mg/dL.
* Proteinuria => 2+ unless all other renal parameters are within normal limits.
* Creatinine clearance < 45 ml/min
* Platelet count less than 130 x 10(3)/microL
* WBC count less than 3.0 x 10(3)/microL
* Patients who are known to be immunosuppressed and/or are receiving chronic immunosuppressive therapy
* Female patients of childbearing potential. Male patients who do not agree to use birth control (condom) for a period of 8 weeks following study product administration
* Investigational drug therapy within 30 days of treatment
* Patients who have received any gene therapy product or angiogenic growth factor protein product
* Underlying disease(s) other than CAD resulting in a life expectancy of less than 1 year
* Any clinical abnormality or social circumstance that puts successful completion of the trial in doubt

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2001-10; Primary Completion 2005-01 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change in treadmill exercise duration from baseline | 12 Weeks

SECONDARY OUTCOMES:
Percentage of patients with a =>30% increase in exercise duration compared to baseline | 4 weeks, 12 weeks and 6 months
Number of patients with and time to coronary events or all-cause death | 1 Year
Change in treadmill exercise duration compared to baseline | 4 weeks and 6 months
Change in time to 1 mm ST segment depression during ETT compared to baseline | 4 weeks, 12 weeks and 6 months
Change in time to angina onset during ETT compared to baseline | 4 weeks, 12 weeks and 6 months
Change in CCS class compared to baseline | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 6 months and 12 months
Change in weekly frequency of anginal attacks compared to baseline | 2 weeks, 4 weeks, 8 weeks, 12 weeks and 6 months
Change in weekly PRN nitroglycerin use compared to baseline | 2 weeks, 4 weeks, 8 weeks, 12 weeks and 6 months
Change in quality of life (SAQ, DASI, SF-36, EQ-5D) compared to baseline | 4 weeks, 12 weeks, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Foster, MD, Study Director — Cardium Therapeutics, 12255 El Camino Real #250, San Diego, CA 92130, (858) 436-1000

REFERENCES:
- [Derived] Henry TD, Grines CL, Watkins MW, Dib N, Barbeau G, Moreadith R, Andrasfay T, Engler RL. Effects of Ad5FGF-4 in patients with angina: an analysis of pooled data from the AGENT-3 and AGENT-4 trials. J Am Coll Cardiol. 2007 Sep 11;50(11):1038-46. doi: 10.1016/j.jacc.2007.06.010. Epub 2007 Aug 24. PMID 17825712